CLINICAL TRIAL: NCT03534076
Title: Predicting Sleep, Smoking, and Lung Health Disparities in African American Adults
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1183509; 1R01MD012734-01 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-05-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Sleep; Lung Diseases; Smoking
MeSH Terms: conditions — Lung Diseases; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cohort Observational study — Cohort Observational study - there is no intervention

SUMMARY:
This 5-year prospective, observational study will: (1) determine the individual, social, and environmental predictors of sleep duration, quality, latency, efficiency, timing and regularity in African American smokers, (2) quantify the prospective relationship between multiple metrics of sleep with tobacco use, such that a sleep phenotype of risk for smoking is defined, and (3) examine the extent to which short sleep (<7 hrs) and other unhealthy sleep metrics, predicts lung function through smoking behaviors and inflammation, in 480 African Americans at risk for advancing COPD (GOLD Stage 0-2 and current smoker). Study subjects will be recruited via Temple Health System sites. Following eligibility screening, initially eligible subjects will provide written study consent and complete an in-home sleep assessment to rule out the exclusionary moderate-severe sleep apnea and other sleep disorders. Consenting and eligible subjects will be entered into the study and across the 60-month data collection period, complete 8 assessments: 4 annual clinical based assessments, interspersed by 4 mid-year, phone-based, self-report assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported African American, White, or mixed ethnicity.
2. 40 - 67 years.
3. GOLD stage 0-3 as assessed by spirometry.
4. No moderate-severe sleep disorders or use of sleep medication.
5. Self-reported current cigarette smoker as defined by smoking one or more cigarettes in the last month.
6. Able to communicate in English and provide written informed consent.

Exclusion Criteria:

1. Self-reported ethnicity (in full or part) other than Black/African American or White.
2. < 40 years of age.
3. Not a current cigarette smoker (< 1 cigarette in last month).
4. GOLD stage >3.
5. Presents with a diagnosed moderate-severe sleep disorder
6. Use of any sleep medication. -

Ages: 40 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population are 480 African American smokers and 80 White smokers who do not have a sleep disorder or GOLD stages 4 at intake.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
FEV1/FVC ratio | 365 days
  Lung function as defined as the ratio of Forced Expiration Volume in one second (FEV1) to the Forced Vital Capacity (FVC; FEV1/FVC ratio) will be computed

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Satti, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Patterson F, Brewer B, Blair R, Grandner MA, Hoopes E, Ma G, Criner GJ, Satti A. An exploration of clinical, behavioral, and community factors associated with sleep duration and efficiency among middle-aged Black/African American smokers. Sleep Health. 2021 Jun;7(3):397-407. doi: 10.1016/j.sleh.2021.01.006. Epub 2021 Mar 16. PMID 33741321
- [Derived] Gangemi AJ, Satti A, Zantah M, Blair R, Brewer B, Ma G, Grandner MA, Davey A, Criner GJ, Patterson F. Sleep Duration and Efficiency Associated With Better Functional Exercise Capacity in Black Smokers at Risk for COPD. Chest. 2020 Oct;158(4):1680-1688. doi: 10.1016/j.chest.2020.03.070. Epub 2020 Apr 22. PMID 32333930